CLINICAL TRIAL: NCT00903799
Title: Clinical Efficacy and Efficiency of Gastric Electrical Stimulation (Enterra®) for Refractory Nausea and/or Vomiting
Brief Title: Medico-economic Evaluation of ENTERRA Therapy
Acronym: ENTERRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2008/046/HP
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Gastroparesis; Vomiting; Nausea
Keywords: Drug-refractory gastroparesis; diabetes mellitus induced gastroparesis; Gastric electrical stimulation; Long-term multicenter study
MeSH Terms: conditions — Gastroparesis; Vomiting; Nausea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Gastric electrical stimulation using Enterra Therapy. Device activated during 4 months then device in 'OFF' position the 4 following months.
  After the cross-over period, device activated until the end of the trial
  Interventions: Device: Implantation of ENTERRA therapy
- 2 (Other): Gastric electrical stimulation using Enterra Therapy. Device in 'OFF' position during 4 months then device activated the 4 following months.
  After the cross-over period, device activated until the end of the trial
  Interventions: Device: Implantation of ENTERRA therapy

INTERVENTIONS:
Device: Implantation of ENTERRA therapy — Gastric electrical stimulation using Enterra Therapy

SUMMARY:
The aim of this clinical trial is to assess the symptomatic efficacy and the impact on the utilization of healthcare resources of a treatment by gastric electrical stimulation (ENTERRA ®) in patients with refractory nausea and/or vomiting leading to a nutritional impairment. Eligible patients will be those with refractory symptoms either idiopathic, postsurgical or due to diabetes mellitus. The duration of the study will be 28 months for each patient.

After a run-in period of 4 months during which a prospective assessment of healthcare resources utilization and of the severity of the symptoms will be obtained, patients will be implanted. The follow-up period after implantation of the device will last 24 months in every patients and will be divided in two parts: a) After the first postoperative month during which the device will remained on the "OFF" position, the first phase of the study will be a randomized double-blind cross-over study with 2 periods of 4 months during which the device will be activated or not. After the 9th month of follow up, the trial will be an open trial and the device will be activated in all patients.

During the whole trial, patients will record all types of healthcare resources utilizations (hospitalizations, drug treatments, endoscopic procedures…) while the symptomatic efficacy of the treatment will be assessed by standard questionnaires at the following visits scheduled at 1, 5, 9, 12, 18, 24 months. The glycemic control will be determined at each visit in diabetic patients. A delayed gastric emptying will not be a selection criteria but we have planned to analyze the clinical results of the treatment in taking into account a delayed or normal gastric emptying during the pre-implantation period. Moreover, gastric emptying studies have been scheduled at 5, 9, 12 and 24 months to test the impact of gastric electrical stimulation on gastric emptying.

ELIGIBILITY:
Inclusion Criteria:

Nausea and/or vomiting refractory to prokinetics and antiemetics fulfilling the following criteria

1. Due to diabetes mellitus type 1, secondary to oesogastric surgery (vagotomy, partial gastric resection) or idiopathic
2. Non related to other cause
3. Chronic (duration > 12 months)
4. Occurring at least weekly
5. Refractory to anti-emetics (chlorpromazine, ondansétron, granisétron) and/or prokinetics (domperidone, metoclopramide, erythromycin),
6. Leading to weight loss or significant reduction of food intake
7. occurring in patients without any contra-indication for the surgical implantation of the device, in particular severe cardiac or respiratory failure or haemostasis disorders,
8. in patients older than 18 years
9. with a negative pregnancy test at entry into the trial in women
10. Patients who signed the study consentment
11. Affiliation to the the welfare system

Exclusion Criteria:

1. Patients older than 70,
2. Patients in whom nausea and/or vomiting are related to another aetiology than that previously described.
3. Patients with an absolute contraindication for general anaethesia and surgery
4. Patients with a contra-indication for implantation of the device
5. Patients with a severe psychiatric disorder
6. Patients under guardianship or curatorship
7. Patients with a major obesity or as severe eating disorder.
8. Patients unable to understand French.
9. Pregnant women or nursing mothers
10. Lack of effective contraception
11. Patients having undergone a pancreatic graft within the previous 6 months and being in a unstable clinical conditions at enrollment
12. Patients with an underlying disease leading to a follow-up by MRI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2009-06; Primary Completion 2014-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
clinical efficacy | 24 months

SECONDARY OUTCOMES:
medico-economic evaluation of ENTERRA therapy | 28 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DUCROTTE, Pr, Principal Investigator — UH Rouen
Locations (21):
- France (21):
  - UH Besancon, Besançon
  - AP-HP Jean Verdier, Bondy
  - UH Bordeaux, Bordeaux
  - UH Clermont Ferrand, Clermont-Ferrand
  - AP-HP Louis Mourier, Colombes
  - Corbeil Essones Hospital, Corbeil-Essonnes
  - UH Grenoble, Grenoble
  - UH Lille, Lille
  - UH Lyon, Lyon
  - UH Marseille, Marseille
  - UH Montpellier, Montpellier
  - UH Nancy, Nancy
  - UH Nantes, Nantes
  - UH Nice, Nice
  - UH Nimes, Nîmes
  - UH Poitiers, Poitiers
  - UH Rennes, Rennes
  - UH Rouen, Rouen
  - UH Strasbourg, Strasbourg
  - UH Toulouse, Toulouse
  - UH Tours, Tours

REFERENCES:
- [Derived] Gourcerol G, Coffin B, Bonaz B, Hanaire H, Bruley Des Varannes S, Zerbib F, Caiazzo R, Grimaud JC, Mion F, Hadjadj S, Valensi P, Vuitton L, Charpentier G, Ropert A, Altwegg R, Pouderoux P, Dorval E, Dapoigny M, Duboc H, Benhamou PY, Schmidt A, Donnadieu N, Ducrotte P, Guerci B; ENTERRA Research Group. Impact of Gastric Electrical Stimulation on Economic Burden of Refractory Vomiting: A French Nationwide Multicentre Study. Clin Gastroenterol Hepatol. 2022 Aug;20(8):1857-1866.e1. doi: 10.1016/j.cgh.2020.11.011. Epub 2020 Nov 13. PMID 33189854
- [Derived] Ducrotte P, Coffin B, Bonaz B, Fontaine S, Bruley Des Varannes S, Zerbib F, Caiazzo R, Grimaud JC, Mion F, Hadjadj S, Valensi PE, Vuitton L, Charpentier G, Ropert A, Altwegg R, Pouderoux P, Dorval E, Dapoigny M, Duboc H, Benhamou PY, Schmidt A, Donnadieu N, Gourcerol G, Guerci B; ENTERRA Research Group. Gastric Electrical Stimulation Reduces Refractory Vomiting in a Randomized Crossover Trial. Gastroenterology. 2020 Feb;158(3):506-514.e2. doi: 10.1053/j.gastro.2019.10.018. Epub 2019 Oct 21. PMID 31647902